CLINICAL TRIAL: NCT06707636
Title: Using Life's Essential 8 to Lower Heart Disease Risk in Midlife Black Women
Brief Title: Using Life's Essential 8 in Midlife Black Women
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Holly Jones, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024B0010
Record Dates: First submitted 2024-11-14; First posted 2024-11-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Stress; Self-Efficacy; Heart Disease Risk Factors; Depression Symptoms; Awareness; Perceived Stress; Lifestyle Intervention; Behavior Change
Keywords: perceived stress; heart disease risk factors; lifestyle intervention; behavior change; strong woman syndrome; choice
MeSH Terms: conditions — Depression | interventions — Health

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black Women's Stress and Wellness (B-SWELL) arm (Experimental): The B-SWELL arm consists of 8-weekly sessions. Sessions last 90 minutes and focus on stress reduction, heart disease, and healthy lifestyle changes. The American Heart Association's Life's Essential 8 metrics are leveraged and culturally tailored in the B-SWELL materials. Participants will also receive personalized health coaching.
  Interventions: Behavioral: Experimental: Black Women's Stress and Wellness (B-SWELL) arm
- Wellness (WE) arm (Active Comparator): This is an attention control group. Participants placed in his arm will receive 8-weekly sessions focused on the Life's Essential 8 metrics. Sessions will last approximately 90 minutes.
  Interventions: Behavioral: Active Comparator: Wellness (WE) arm

INTERVENTIONS:
Behavioral: Experimental: Black Women's Stress and Wellness (B-SWELL) arm — The B-SWELL arm consists of 8-weekly sessions. Sessions last 90 minutes and focus on stress reduction, heart disease, and healthy lifestyle changes. The American Heart Association's Life's Essential 8 metrics are leveraged and culturally tailored in the B-SWELL materials. Participants will also receive personalized health coaching.
  Arms: Black Women's Stress and Wellness (B-SWELL) arm
Behavioral: Active Comparator: Wellness (WE) arm — This is an attention control group. Participants placed in his arm will receive 8-weekly sessions focused on the Life's Essential 8 metrics.
  Arms: Wellness (WE) arm

SUMMARY:
This research seeks to improve the Midlife Black Women's Stress Reduction and Wellness Intervention (B-SWELL), a program designed to lower heart disease risk in midlife Black women. The B-SWELL leverages stress reduction to facilitate the adoption and adherence to healthier lifestyle behaviors. This research study will use choice to increase engagement and minimize the effect of social determinants of health on research participation among midlife Black women.

A comparative clinical trial will be conducted. Midlife Black women (ages 45-64) who reside in the Greater Cincinnati area will be recruited for participation. Women are eligible if they self-identify as Black/ African American, are between the ages of 45-64, and are willing to commit to the requirements of the study (e.g., attend 8 weekly sessions and 4 phone interviews). Participants will be randomly placed (like the flip of a coin) into either the B-SWELL or WE group. Both the B-SWELL and WE groups are 8-week programs that focus on healthy lifestyle behaviors and heart disease awareness. Women will have the choice to participate in person or virtually. Survey phone interviews will be conducted at baseline, 8-, 12-, and 16-weeks. Data collected will provide information about adherence, healthy lifestyle behaviors, and cardiovascular health. Heart health will be measured using the American Heart Association's Life's Essential 8 metric.

Outcome measures include heart disease awareness, Life's Essential 8 score, stress, self-efficacy, depressive symptoms, and symptoms.

DETAILED DESCRIPTION:
Conduct a RCT pilot of the modified B-SWELL consisting of 64 women randomized to B-SWELL (n=32) or control (n=32). The RCT will take place in two phases. Each phase will consist of virtual and in-person groups (n=8 for groups) for the B-SWELL and attention control. Participants will receive the B-SWELL materials (binder, flash drive) prior to start. Each weekly 90-minute session is devoted to a specific LE8 behavior. Sessions will begin with meditative practice followed by interactive presentations, review of case studies, and discussion. Coaching will occur via phone during the first weeks of the intervention with booster sessions at weeks 10 and 14. The attention control (virtual or in person) will mirror the B-SWELL in format and duration however, participants will only receive publicly available AHA materials and information. The Attention control will not receive stress information, goal setting, or coaching. Facilitators and coaches will be purposefully recruited and representative of midlife Black women.

This study will take place in Cincinnati. Women will be eligible if they identify as Black/African American; are between the ages of 45 and 64 during the trial; have a reliable phone for messaging and data collection calls; and willing to commit to the study duration and data collection phone calls (at 8, 12 and 16 weeks). Women will be excluded if they have recently immigrated or resettled in the U.S. or have major health conditions prohibiting safe participation. Having CVD will not be an exclusion as those with CVD can still show improvement in LE8. Recruitment activities will include fliers, email, snowballing, and social media. Community in-person sites will be selected based upon safety, accessibility, and resources. The C-RAB members will inform recruitment through their knowledge of the communities. For example, they may recommend that fliers be placed in particular high-traffic areas or sent to specific community organizations. C-RAB members are not personnel and, thus, will be instructed to refer any questions regarding this research to the PI and/or research staff. All C-RAB activities will be monitored by the PI.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as Black/ African American
* Age 45-64.
* Willing to adhere to the study requirements.

Exclusion Criteria:

* Incarcerated or on house arrest,
* Diagnosed with terminal illness, severe mental illness, or dementia.
* Unable or unwilling to participate in 8 weekly sessions and 4 phone interviews.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Life's Essential 8 (LE8) score | From baseline to 16 weeks
  Life's Essential 8 (LE8) is a recognized metric for cardiovascular health as defined by the American Heart Association. The LE8 score consists of 8 sub-measures. There are 4 lifestyle behaviors (Diet, Physical Activity, Nicotine Exposure and Sleep Health) and 4 health factors (BMI, Blood Lipids, Blood Glucose, and Blood Pressure). The total LE8 score is calculated as the average of the 8 individual component scores. Total scores range from 0 to 100 points. Higher scores correspond to better cardiovascular health.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | from baseline to 16 weeks.
  Diagnostic instrument for depression symptoms. The PHQ-9 scores each of the 9 DSM-IV criteria. Question 9 screens for the presence of suicide ideation. Total scores greater than 15 are associated with moderately severe and severe depression.
Pittsburgh Sleep Quality Index (PSQI) | From baseline to 16 weeks
  19-item self-report assessment of sleep quality for the previous 1-month period. Yields 7 sleep components. Each component score ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
researcher-developed symptoms check list | From baseline to 16 weeks
  Participants self-report symptoms experienced over previous 2 weeks in the checklist. Responses are yes/no.

OTHER OUTCOMES:
Perceived stress (PSS-10) | from baseline to 16 weeks.
  Measures perception of general stress. Items rated on a scale of 0-4. Higher scores correspond with higher stress.
Genral Self Efficacy (GSE) | From baseline to 16 weeks
  10-item psychometric scale assesses optimistic self-beliefs to cope with life demands. Each item is scored from 1 (not true) to 4 (exactly true). Higher scores correspond with higher self efficacy.
Super Woman Syndrome | baseline
  cultural constructs related to strength, emotional suppression, vulnerability, motivation, and obligation. Sub scores are summed. Higher scores represent greater endorsement of each item.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will provide prospective survey data from a randomized pilot trial at four timepoints over a period of 16 weeks. The sample (N=64) consists of Black women ages 45-64.
  The data collected will include survey responses designed to assess viability of the optimized Midlife Black Women's Stress and Wellness intervention (B-SWELL). Surveys will include researcher developed tools (i.e., demographics, satisfaction, feedback, and symptoms check list), and seven validated tools (Cohen's Perceived Stress Scale, General Self-Efficacy scale, American Heart Association's Life's Essential 8 score, Perceived General Health scale, Patient Health Questionnaire, and Pittsburgh Sleep Quality Index). Coding, recodes, and analyses related to each tool will be performed according to instruction as they have been validated to ensure production of accurate results.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be will placed in the generalist database, DRYAD in accordance with NIH recommendations, at the time of publication. Data will then remain in DRYAD in perpetuity.
Access Criteria: Studies registered in Dryad are assigned a citable digital object identifier (DOI) number. Studies can be searched by name, DOI identifier, or topic. Datasets in DRYAD are indexed by the Thomson-Reuters Data Citation Index and include schema.org mark-up to make them discoverable in Google Dataset Search. DRYAD also integrates with any SWORD/OAI-PMH compliant repository, allowing its records to be discoverable through additional third-party aggregators.
URL: https://datadryad.org/stash